CLINICAL TRIAL: NCT05634148
Title: Effect of a Single Dose Infusion of Dexmedetomidine in Reducing Incidence of Emergence Agitation After Nasal Surgery - a Randomised Contolled Trial
Brief Title: Dexmedetomidine in Reducing Incidence of Emergence Agitation After Nasal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, Anwar ul Huda, Principle Investigator, Security Forces Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SFH-Dex Nasal
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patients in this group will receive intravenous dexmedetomidine before extubation
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Patients in this group will receive intravenous placebo (0.9 % saline) before extubation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous dexmedetomidine will be administered 45 minutes before extubation in intervention group
  Other Names: Control

SUMMARY:
Various pharmacological interventions have been attempted previously to prevent postoperative EA with variable results. These include use of opioids, propofol, midazolam, ketamine, magnesium and alpha-2 agonists like clonidine and dexmedetomidine. Dexmedetomidine have been used with different dosages and different timings of administration with variable results and at the expense of major hemodynamic disturbances. The objective of this study was to investigate the role of single dose of dexmedetomidine (0.5 mcg/kg) administered as 30 minutes infusion prior to extubation in reducing the incidence and severity of EA and coughing on extubation.

DETAILED DESCRIPTION:
Emergence agitation (EA) or delirium is a post anesthesia complication which is manifested as confusion, agitation, disorientation and aggressive behavior. It can lead to serious consequences including hemorrhage, removal of lines, drains and catheters, self-extubation and even falling out of bed resulting in severe injuries. EA is associated with cognitive deficit, physical dependence, increased hospital stay and higher mortality.

There is wide variation in the incidence of EA in scientific literature ranging from 5 % to 27.3 %. There are no clear diagnostic criteria for EA because of its varied clinical manifestations. Although many risk factors have been identified including pain, presence of stress at the time of induction, induction with etomidate, use of premedication with benzodiazepines, hypoxemia, type of surgery, awakening in hostile and noisy environment and presence of urinary catheter. Patients undergoing nasal surgeries are in particular, at higher risk for EA due to a sense of suffocation secondary to nasal packing.

Various pharmacological interventions have been attempted previously to prevent postoperative EA with variable results. These include use of opioids, propofol, midazolam, ketamine, magnesium and alpha-2 agonists like clonidine and dexmedetomidine. Dexmedetomidine have been used with different dosages and different timings of administration with variable results and at the expense of major hemodynamic disturbances. The objective of this study was to investigate the role of single dose of dexmedetomidine (0.5 mcg/kg) administered as 30 minutes infusion prior to extubation in reducing the incidence and severity of EA and coughing on extubation.

ELIGIBILITY:
Inclusion Criteria:

* We will include patients aged 15 years to 65 years, ASA 1-3 who are planned to undergo general anesthesia for elective nasal surgeries in which nasal packing is used postoperatively

Exclusion Criteria:

* We will exclude patients with known allergy to study medications, BMI more than 35, history of obstructive sleep apnea, history of psychiatric illness, pregnancy and presence of liver and renal diseases.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Riker sedation-agitation score | 60 minutes
  Assessment of emergence delirium after extubation. It has numbers from 1-7.

SECONDARY OUTCOMES:
Postoperative pain score | 60 minutes
  Numerical rating scale pain score in PACU. from 0 to 10 with 10 worst pain
Opioid consumption | 60 minutes
  Morphine equivalent consumption in PACU
Adverse events | 60 minutes
  Intraoperative or postoperative adverse events
Duration of stay in PACU | 60 minutes
  duration of PACU stay

CONTACTS AND LOCATIONS:
Overall Officials: Anwar Huda, FRCA, Principal Investigator — Security Forces Hospital
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR